CLINICAL TRIAL: NCT02635607
Title: A RCT Study to Evaluate the Safety and Efficacy of the Fixed Day-5 Antagonist Protocol Versus the Flexible Antagonist Protocol for the Controlled Ovarian Stimulation in Chinese Women With Predicted High Ovarian Response
Brief Title: Effectiveness and Safety Study of Fixed Versus Flexible of Gonadotropin-releasing Hormone Antagonist Protocol
Acronym: GnRH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chong Qing Reproducive and Genetic Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Merck-IISP-01
Record Dates: First submitted 2015-12-11; First posted 2015-12-21 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-12

CONDITIONS: Infertility
Keywords: GnRH antagonist; fixed protocol; flexible protocol
MeSH Terms: conditions — Infertility | interventions — follitropin beta; ganirelix; Ovidrel; Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fixed Protocol (Other): Patients will start Follitropin beta stimulation on menstrual cycle day 3 and the daily dose will be fixed for the first 5 days of stimulation, a modification of the rFSH dose will be allowed from stimulation day 6 onward. Ganirelix will start fixedly on stimulation Day 5. rhCG will be administered to induce final oocyte maturation as soon as at least three follicles of ≥17 mm were observed, and triptorelin trigger will be used as a replacement in case of OHSS high risk
  Interventions: Drug: Follitropin Beta; Drug: Ganirelix; Drug: rhCG; Drug: triptorelin
- Flexible protocol (Other): Patients will start Follitropin beta stimulation on menstrual cycle day 3 and the daily dose will be fixed for the first 5 days of stimulation, a modification of the rFSH dose will be allowed from stimulation day 6 onward. Ganirelix will start flexibly by the promissory criterion in the flexible group. rhCG will be administered to induce final oocyte maturation as soon as at least three follicles of ≥17 mm were observed, and triptorelin trigger will be used as a replacement in case of OHSS high risk
  Interventions: Drug: Follitropin Beta; Drug: Ganirelix; Drug: rhCG; Drug: triptorelin

INTERVENTIONS:
Drug: Follitropin Beta — Patients will start stimulation with a daily s.c. injection of 150IU follitropin beta on menstrual cycle day 3. A modification of the rFSH dose will be allowed from stimulation day 6 onward in case that a high ovarian response occurs at the discretion of the investigator.
  Other Names: Puregon
Drug: Ganirelix — Ganirelix 0.25mg daily s.c. will start after 4 days of rFSH stimulation
  Other Names: Orgalutran
  Arms: Fixed Protocol
Drug: Ganirelix — Ganirelix 0.25mg daily s.c. will start when at least one of the following criteria are fulfilled: (i) the presence of at least one follicle measuring≥12 mm; (ii) serum E2 levels>600 pg/ml; and (iii) serum LH levels>10 IU/l.
  Other Names: Orgalutran
  Arms: Flexible protocol
Drug: rhCG — An amount of 250ug rhCG will be administered to induce final oocyte maturation as soon as at least three follicles of ≥17 mm were observed
  Other Names: Ovidrel
Drug: triptorelin — 0.2mg triptorelin will replace rHCG to trigger in case of high risk of overstimulation
  Other Names: Decapeptyl

SUMMARY:
The purpose of study is to compare the effectiveness of the Day-5 fixed administration of GnRH antagonist versus flexible administration of GnRH antagonist during ovarian stimulation in Chinese women with predicted high ovarian response, and the hypotheses is that the number of oocyte retrieved in fixed protocol is not inferior to GnRH antagonist flexible protocol.

DETAILED DESCRIPTION:
The investigator will be responsible for analyzing the study data. This study is designed as an open-label fashion, and thus, no blindness will be maintained during the study. The database will not be locked until medical/scientific review has been completed, protocol violators have been identified, and data has been declared complete.

Statistical Methods For the primary endpoint, mean and standard deviation (SD) on the number of oocytes will be presented. The between-group difference and corresponding 95% confidence interval (CI) (Day-5 fixed protocol - flexible protocol) will be calculated by using a two-sample t-test under the assumption that the sample data are normally distributed. A test for normality will be performed prior to the analysis on primary endpoint and possible nonparametric adjustment will be made for skewed data in terms of primary analyses. The non-inferiority will be established if the lower bound of the 95%CI in the treatment difference between two groups (Day-5 fixed protocol - flexible protocol) does not exceed -3.0. The superiority may be claimed for the Day-5 fixed protocol if the lower bound of 95%CI for the treatment difference is above 0.0.

For the secondary endpoints on categorical variables, the number and percentage of the event will be calculated and displayed. Clinical and ongoing pregnancy rates will be separately calculated and presented. Between-group comparisons will be made by Chi-square test and the corresponding 95%CI will be presented by using Miettinen-Nurminen method if the number of the observed events is at least 4. Mean and SD will be summarized for continuous variables in terms of secondary outcome measures. A treatment difference between study groups will be made by using two-sample t-test or nonparametric test whenever appropriate.

The number of subjects who have reported adverse experiences (AE) and the incidence of individual AEs will be counted and presented. Fisher's exact test will be performed to compare between treatment groups.

Demographics and the subject's relevant medical history will be summarized by descriptive statistics.

All statistical analyses will be two-sided and at a significant level of a p value less than 0.05, unless otherwise specified.

Sample Size:

A sample size of 200 (1:1 allocation) achieves 80% power to detect non-inferiority of the Day-5 fixed-dose regimen as compared with the flexible protocol by a margin at -3 oocytes retrieved (3 oocytes fewer than the controlled group), using a one-sided, two-sample t-test with Mann-Whitney test adjustment at the significance level at 0.025. The true difference between the means is assumed to be 0.0 and the standard deviation of both intervention arms to be 6.8. The pre-mature discontinuation rate is set at approximately 15% for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Have an indication for COS and IVF/ICSI;
2. be <35 years old;
3. have a BMI of 18-25kg/m2;
4. have a regular menstruation with a range of 24-35 days;
5. fulfill one of these three criteria as follow:

   * the number of oocytes retrieved>15 in previous COS cycle;
   * Serum AMH (examined on the menstrual cycle day 2)>3.52ng/ml;
   * antral follicle count (AFC) (examined by ultrasonic on the menstrual cycle day 2)>16
6. have willingness to give informed consent

Exclusion Criteria:

1. Presence of unilateral ovary absence;
2. Any difficulty on oocyte pick-up with abnormal condition of ovary and pelvic cavity;
3. Women have any clinically relevant pathology could impair embryo implantation or pregnancy continuation (uterine malformation, intermural uterine fibroids>3cm, intrauterine adhesion,etc);
4. Women with polycystic ovary syndrome (PCOS) diagnosed by Rotterdam consensus criterion(Rotterdam, 2004)
5. Other known abnormal ovulation disorders (including but not limited to adrenal gland disease, thyroid disease and hyperprolactinemia);
6. A history of recurrent miscarriage or previous IVF cycles failure>2;
7. A history of ovarian hypo-response in previous ovarian stimulation;
8. Women with other clinical/socio-economic factors precluding the completion of the study at the discretion of the investigator.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
the number of oocytes retrieved | 3 weeks

SECONDARY OUTCOMES:
Total dosage of Gn and GnRH antagonist | 3 weeks
The incidence of premature LH surge during the stimulation | 3 weeks
The incidence of OHSS during the study | 5 weeks
The implantation rate | 5 weeks
  the implantation rate is defined as the number of gestational sac observed by ultrasound examination at 4 weeks after ET per 100 embryos transferred
clinical pregnancy rate | 6 weeks
  Clinical pregnancy was defined as the presence of a gestation sac with a positive heartbeat detectable by transvaginal ultrasonography at 6 weeks after ET.
ongoing pregnancy rate | 14 weeks
  Ongoing pregnancy was defined as a pregnancy with cardiac activity proceeding beyond 12 weeks of gestation.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Ye, bachelor, Study Director — Genetic and Reproductive Institute, Chongqing Obstetrics and Gynecology Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Humaidan P, Quartarolo J, Papanikolaou EG. Preventing ovarian hyperstimulation syndrome: guidance for the clinician. Fertil Steril. 2010 Jul;94(2):389-400. doi: 10.1016/j.fertnstert.2010.03.028. Epub 2010 Apr 22. PMID 20416867
- [Background] Al-Inany HG, Youssef MA, Aboulghar M, Broekmans F, Sterrenburg M, Smit J, Abou-Setta AM. Gonadotrophin-releasing hormone antagonists for assisted reproductive technology. Cochrane Database Syst Rev. 2011 May 11;(5):CD001750. doi: 10.1002/14651858.CD001750.pub3. PMID 21563131
- [Background] Lainas TG, Sfontouris IA, Zorzovilis IZ, Petsas GK, Lainas GT, Alexopoulou E, Kolibianakis EM. Flexible GnRH antagonist protocol versus GnRH agonist long protocol in patients with polycystic ovary syndrome treated for IVF: a prospective randomised controlled trial (RCT). Hum Reprod. 2010 Mar;25(3):683-9. doi: 10.1093/humrep/dep436. Epub 2009 Dec 15. PMID 20008886
- [Background] Al-Inany H, Aboulghar MA, Mansour RT, Serour GI. Optimizing GnRH antagonist administration: meta-analysis of fixed versus flexible protocol. Reprod Biomed Online. 2005 May;10(5):567-70. doi: 10.1016/s1472-6483(10)61661-6. PMID 15949209
- [Background] Hamdine O, Eijkemans MJ, Lentjes EW, Torrance HL, Macklon NS, Fauser BC, Broekmans FJ. Ovarian response prediction in GnRH antagonist treatment for IVF using anti-Mullerian hormone. Hum Reprod. 2015 Jan;30(1):170-8. doi: 10.1093/humrep/deu266. Epub 2014 Oct 29. PMID 25355590
- [Background] Engmann L, DiLuigi A, Schmidt D, Nulsen J, Maier D, Benadiva C. The use of gonadotropin-releasing hormone (GnRH) agonist to induce oocyte maturation after cotreatment with GnRH antagonist in high-risk patients undergoing in vitro fertilization prevents the risk of ovarian hyperstimulation syndrome: a prospective randomized controlled study. Fertil Steril. 2008 Jan;89(1):84-91. doi: 10.1016/j.fertnstert.2007.02.002. Epub 2007 Apr 26. PMID 17462639
- [Derived] Luo X, Pei L, Li F, Li C, Huang G, Ye H. Fixed versus flexible antagonist protocol in women with predicted high ovarian response except PCOS: a randomized controlled trial. BMC Pregnancy Childbirth. 2021 May 2;21(1):348. doi: 10.1186/s12884-021-03833-2. PMID 33934703